CLINICAL TRIAL: NCT02839382
Title: The Northwest Coalition for Primary Care Practice Support
Acronym: H2N
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: University of Washington (Other); Oregon Health and Science University (Other); Qualis Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: AHRQ 1R8HS023908-01
Record Dates: First submitted 2016-07-18; First posted 2016-07-21 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Cardiovascular Disease; Essential Hypertension; Nicotine Dependence; Hyperlipidemia
MeSH Terms: conditions — Cardiovascular Diseases; Essential Hypertension; Tobacco Use Disorder; Hyperlipidemias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Coaching (Active Comparator): External facilitation by a practice coach for 15 months
  Interventions: Other: Coaching
- Educational Outreach (Active Comparator): Academic detailing phone calls to support implementation of a cardiovascular risk calculator/estimator in each clinic
  Interventions: Other: Coaching; Other: Educational Outreach
- Site Visit (Active Comparator): Site visits made by practices to 'exemplar" practices to learn innovative approaches to quality improvement
  Interventions: Other: Coaching; Other: Site Visits
- Educational Outreach and Site Visit (Active Comparator): In this arm of the study, practices will be offered both educational outreach and an opportunity for a site visit
  Interventions: Other: Coaching; Other: Educational Outreach; Other: Site Visits

INTERVENTIONS:
Other: Coaching — An external facilitator or coach is assigned 15-20 primary care clinics and will make face-to-face site visits and monthly phone calls for 15 months to support building QI capacity in each assigned practcie
  Other Names: Practice Facilitation
Other: Educational Outreach — Practices randomized to this arm of the study will receive an educational outreach phone call by an academic expert on implementation strategies for use of a cardiovascular risk calculator within their daily work flow and clinic setting
  Other Names: Academic Detailing
  Arms: Educational Outreach; Educational Outreach and Site Visit
Other: Site Visits — Practices randomized to this arm of the study will be given an opportunity to make a site visit to an "exemplar" practice to learn about innovative approaches to conducting quality improvement activities.
  Other Names: Peer-to-peer learning
  Arms: Educational Outreach and Site Visit; Site Visit

SUMMARY:
The purpose of this project is to build capacity for quality improvement (QI) in small primary care practices across Washington, Oregon and Idaho by improving risk factors for heart attacks such as blood pressure, cholesterol and smoking. The Northwest Coalition for Primary Care Practice Support will assist practices by providing them with a QI coach, creating group learning opportunities, and conducting educational outreach activities. An innovative study design will be used to determine what levels and types of support are most helpful and effective.

DETAILED DESCRIPTION:
The Northwest Coalition for Primary Care Practice Support will provide a comprehensive and robust external practice support infrastructure for small and medium primary care practices across Washington (WA), Oregon (OR) and Idaho (ID) to build their internal quality improvement (QI) capacity and improve performance on the heart health indicators of aspirin use, blood pressure and cholesterol control and smoking cessation (ABCS indicators) by disseminating and supporting the implementation of relevant Patient Centered Outcomes Research findings. This coalition of partners has a remarkable track record of collaboration and improving primary care practice: the MacColl Center for Health Care Innovation and the Center for Community Health Evaluation at Group Health Research Institute; Qualis Health, the Health IT Regional Extension Center (REC) and designated Quality Improvement Organization (QIO) for WA and ID; and the Oregon Rural Practice-based Research Network (ORPRN), along with state-level partners who are membership organizations for clinicians in small practice settings. Recruitment will leverage existing small practice relationships between Qualis Health as the health information technology (IT) REC for WA and ID and ORPRN's existing network of small practices with a goal of enrolling 320 small practices out of an estimated 1,479 with stage 1 meaningful use of their electronic health record across the three states. In addition to providing health IT support for the Physician Quality Reporting System (PQRS) to measure the ABCS indicators in all practices, our comprehensive approach to building QI capacity and improving the ABCS measures consists of: 1) practice facilitation as a unifying strategy, 2) academic detailing/outreach to support implementation of PCOR findings, and 3) shared learning collaboratives. We will employ an innovative study and evaluation design by providing two levels of support for each of the latter three practice support components. By randomly assigning practices to one of eight possible combinations of practice support, we will "…develop new evidence about the contribution of various components of the comprehensive approach and the effect of the intensity of the approach on outcomes." Our rigorous mixed-method evaluation is based on the RE-AIM framework and will employ multi-level models and interrupted time series regression. Data will be collected from a control group of practices to examine secular trends. Our Specific Aims are to: 1) Identify, recruit and conduct baseline assessments in 320 small to medium size primary care practices across the geographically contiguous region of WA, OR and ID; 2) Provide comprehensive external practice support to build QI capacity within these practices; 3) Disseminate and support the adoption of PCOR findings relevant to the ABCS quality measures; 4) Conduct a rigorous evaluation of the effectiveness of providing external practice support to implement PCOR findings and improve ABCS measures; and 5) Assess the sustainability of changes made in QI capacity and ABCS improvements and develop a model of dissemination and primary care practice support infrastructure.

ELIGIBILITY:
Inclusion Criteria:

* Primary care practice with 10 or fewer providers and an Electronic Health Record (EHR) that meets Stage 1 meaningful use criteria

Exclusion Criteria:

* No EHR

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Appropriate use of Aspirin | Every 3 months with 12 month look-back
  National Quality Forum (NQF) 0068 Ischemic Vascular Disease (IVD): Use of Aspirin or another Antithrombotic
Hypertension | Every 3 months with 12 month look-back
  NQF 0018 Controlling hypertension
Smoking | Every 3 months with 12 month look-back
  NQF 0027 Smoking and Tobacco Use Cessation, Medical Assistance

SECONDARY OUTCOMES:
Change Process Capacity | Baseline, 15 months, 21 months
  The change process capacity questionnaire
Quality Improvement Capacity Assessment | Baseline and 12 months
  Practice-level consensus agreement on QI capacity

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Parchman, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- GroupHealthCoop, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Parchman ML, Fagnan LJ, Dorr DA, Evans P, Cook AJ, Penfold RB, Hsu C, Cheadle A, Baldwin LM, Tuzzio L. Study protocol for "Healthy Hearts Northwest": a 2 x 2 randomized factorial trial to build quality improvement capacity in primary care. Implement Sci. 2016 Oct 13;11(1):138. doi: 10.1186/s13012-016-0502-7. PMID 27737719
- [Background] Fagnan LJ, Walunas TL, Parchman ML, Dickinson CL, Murphy KM, Howell R, Jackson KL, Madden MB, Ciesla JR, Mazurek KD, Kho AN, Solberg LI. Engaging Primary Care Practices in Studies of Improvement: Did You Budget Enough for Practice Recruitment? Ann Fam Med. 2018 Apr;16(Suppl 1):S72-S79. doi: 10.1370/afm.2199. PMID 29632229
- [Background] Baldwin LM, Fischer MA, Powell J, Holden E, Tuzzio L, Fagnan LJ, Hummel J, Parchman ML. Virtual Educational Outreach Intervention in Primary Care Based on the Principles of Academic Detailing. J Contin Educ Health Prof. 2018 Fall;38(4):269-275. doi: 10.1097/CEH.0000000000000224. No abstract available. PMID 30346338
- [Derived] Tuzzio L, O'Meara ES, Holden E, Parchman ML, Ralston JD, Powell JA, Baldwin LM. Barriers to Implementing Cardiovascular Risk Calculation in Primary Care: Alignment With the Consolidated Framework for Implementation Research. Am J Prev Med. 2021 Feb;60(2):250-257. doi: 10.1016/j.amepre.2020.07.027. Epub 2020 Dec 3. PMID 33279368
- [Derived] Parchman ML, Anderson ML, Penfold RB, Kuo E, Dorr DA. The Ability of Practices to Report Clinical Quality Measures: More Evidence of the Size Paradox? J Am Board Fam Med. 2020 Jul-Aug;33(4):620-625. doi: 10.3122/jabfm.2020.04.190369. PMID 32675274
- [Derived] Parchman ML, Anderson ML, Coleman K, Michaels LA, Schuttner L, Conway C, Hsu C, Fagnan LJ. Assessing quality improvement capacity in primary care practices. BMC Fam Pract. 2019 Jul 25;20(1):103. doi: 10.1186/s12875-019-1000-1. PMID 31345167